CLINICAL TRIAL: NCT03166202
Title: Age-Related Macular Degeneration, Scotopic Dysfunction, and Driving Performance in a Simulator
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Cynthia Owsley, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 228382017
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous work collectively suggests that rod-mediated dark adaptation (RMDA) is a promising candidate as a functional endpoint measure for evaluating interventions to slow early progression of age-related macular degeneration (AMD). However, there is no agreement among the clinical, research and regulatory communities as to what constitutes a clinically (practically) significant slowing in RMDA. Treatments for AMD are often not considered efficacious if they do not result in a criterion level of improvement in vision. But how much change in the rate of dark adaptation constitutes a clinically significant change? Until this issue is resolved, progress in developing clinical trials on early AMD are at a standstill since there is no functional endpoint to be used in the trial. One approach to establishing clinical significance is to examine how RMDA relates to the performance of an everyday visual task under low luminance conditions, such as night driving or reading. However, such data are not yet available. The purpose of this project is to examine the relationship between RMDA and night-time driving and reading under poor illumination. This information will guide the development of a definition of a clinically significant difference in RMDA that can be used in designing clinical trials on early AMD.

DETAILED DESCRIPTION:
The specific aims of this study are as follows:

Aim 1: To examine the association between RMDA as assessed by the rod intercept time and self reported driving difficulty and experiences during night time driving.

Aim 2: To examine the association between RMDA as assessed by rod intercept time and reading performance as assessed by the MNREAD test administered under a low light level. Reading performance will be defined in terms of maximum reading speed, critical print size (i.e., the smallest print size that supports maximum reading speed), reading acuity (i.e., the smallest print size that can be just read) and the reading accessibility index (i.e., an individual's access to text over the range of print sizes found in everyday life).

ELIGIBILITY:
Inclusion Criteria:

* age-related macular degeneration in one or both eyes, ability to follow simple instructions, licensed to drive a vehicle, can read and speak English

Exclusion Criteria:

* diabetes, retinal or optic nerve conditions other than age-related macular degeneration, neurological conditions that impair vision

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living in the community who have current driver's license who have age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
rod intercept time | measured once (1 day)
  rate of rod-mediated dark adaptation

SECONDARY OUTCOMES:
severity of age-related macular degeneration | measured once (1 day)
  defined by grading of color fundus photos

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owsley, PhD, Principal Investigator — University of Alabama at Birmingham; MiYoung Kwon, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Callahan Eye Hospital, UAB Dept of Ophthalmolog & Visual Sciences, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once study is completed and published in the peer review literature, we will arrange for a data sharing process with other researchers

REFERENCES:
- [Background] Owsley C, McGwin G Jr, Clark ME, Jackson GR, Callahan MA, Kline LB, Witherspoon CD, Curcio CA. Delayed Rod-Mediated Dark Adaptation Is a Functional Biomarker for Incident Early Age-Related Macular Degeneration. Ophthalmology. 2016 Feb;123(2):344-351. doi: 10.1016/j.ophtha.2015.09.041. Epub 2015 Oct 30. PMID 26522707